CLINICAL TRIAL: NCT00392249
Title: Supervised Treatment in Outpatients for Schizophrenia (STOPS)Versus Treatment as Usual in Outpatients, a Randomized Controlled Trial.
Brief Title: Supervised Treatment of Schizophrenia, a Randomized Controlled Trial.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lady Reading Hospital, Pakistan (Other Government)
Collaborators: GTZ Pakistan (German Technical Cooperation) (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGMILRH 01
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2008-02-27 (Estimated); Status verified 2008-02

CONDITIONS: Schizophrenia; Schizoaffective Disorders
Keywords: Schizophrenia; Drug adherence
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Medication Adherence

INTERVENTIONS:
Behavioral: Supervised Treatment of Schizophrenia by a family member

SUMMARY:
Patients suffering from Schizophrenia and their families often suffer from poor care because of ignorance about the disorder especially in economically developing countries. Although antipsychotic medication is effective in reducing relapse rate, 30-40 percent of patients relapse within one year and 40-60 percent relapse within 2 years after discharge from 1st hospitalization even if they are receiving maintenance medication.

Although antipsychotic medications are the mainstay of the treatment for schizophrenia, patients with schizophrenia benefit more from combined use of antipsychotic drugs and psychosocial treatment than pharmacotherapy alone in delaying or preventing relapse or reducing hospital days. It is also less costly than standard treatment and suitable for psychiatric rehabilitation.

Although there are now a number of studies from western countries and a randomized controlled trial from china which have led to increase enthusiasm about psychosocial treatment for schizophrenia but question remains about comparative benefit of treatment methods and additional methods of multiple treatment. In developing countries there is need for further studies in which integrated treatment of pharmaco-therapy and psycho-education is instituted and compared with treatment as usual.

Realizing the need for maintaining the compliance and continuity of treatment, department of psychiatry has started a program called Supervised Treatment of Outpatient Schizophrenia. This study aims to evaluate the effectiveness of Supervised Treatment versus the usual care provided in the outpatient.

DETAILED DESCRIPTION:
Introduction:

Schizophrenic patients and their families often suffer from poor care because of ignorance about the disorder1, especially in economically developing countries. Although many patients of schizophrenia respond well to antipsychotic treatment, the risk of subsequent relapses is generally high2, 40-60 percent relapse within 2 years after discharge from 1st hospitalization is observed even if they are receiving maintenance medication1.

Also non-compliance is quite common in patients with schizophrenia like any other illness, and it should be addressed3 because noncompliance and aggression risk profile symptoms are positively correlated to hospitalization4.

Non-compliance is also common in Pakistan like any other society. The commonest reasons for non-compliance are unawareness of the benefits of treatment, non affordability of drugs, physical side effects, no awareness given by the doctor and unfriendly attitude of doctors5.

Educational therapy both for patient and family led to significant psychopathological improvement at post-treatment and at follow-up.6 The recent trend of family intervention produced many models. One long-term family based intervention reduced the risk of psychotic relapse to about the half within the first two years. These methods also shorten hospital stays, improve compliance with medication, patients' social functioning and relatives' well-being, and they seem to be cost-effective.7 Definitive relationship exists between compliance and the economic costs of schizophrenia as lower rates of compliance lead to higher costs of treating schizophrenia8.

Family education on schizophrenia in China was effective in improving knowledge and promoting improvement in patients' symptoms9. A largest randomized controlled trial from china10 have led to increase enthusiasm about psychosocial treatment for schizophrenia but question remains about comparative benefit of treatment methods and additional methods of multiple treatment11.

Mostly research done on role of psychosocial-education in schizophrenia is from developed countries but no work has been done yet in developing country like Pakistan even Subcontinent having a different cultural background. Realizing the need for maintaining the compliance and continuity of treatment, I have designed a study program called Supervised Treatment of Outpatient Schizophrenia. This study aims to evaluate the effectiveness of Supervised Treatment versus the usual care provided in the outpatient.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia or schizoaffective disorder based on the ICD-10 criteria for schizophrenia.
2. Patients requiring treatment in outpatients
3. Residence in Peshawar district
4. Patient living with relative(care giver) for at least six months.

Exclusion Criteria:

1. Evidence of organic mental disorder
2. Evidence of mental retardation
3. Severe drug dependence requiring inpatient treatment and/or detoxification

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-09 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
To compare the compliance in patients suffering from schizophrenia with Supervised Treatment in Outpatients for Schizophrenia with Treatment As Usual (TAU, control group)

SECONDARY OUTCOMES:
To compare the effectiveness of Supervised Treatment in Outpatients of Schizophrenia with Treatment As Usual (TAU, control group) in preventing relapse and rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Farooq, MCPS,FCPS, Principal Investigator — • Associate Professor, and Head Department of Psychiatry, Postgraduate Medical Institute, (P.G.M.I) Hayat Abad Medical Complex, Peshawar, Pakistan and consultant Psychiatrist Lady Reading Hospital, Peshawar. Pakistan
Locations (1):
- Department of Psychiatry, Peshawar, Khyber Pakhtunkhwa, Pakistan